CLINICAL TRIAL: NCT00625664
Title: Randomized Study of LAROTAXEL + Cisplatin (LC) vs. Gemcitabine + Cisplatin (GC) in the First Line Treatment of Locally Advanced/Metastatic Urothelial Tract or Bladder Cancer
Brief Title: Larotaxel + Cisplatin Versus Gemcitabine + Cisplatin in First Line Treatment of Locally Advanced/Metastatic Urothelial Tract or Bladder Cancer
Acronym: CILAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6668; EUDRACT: 2007-001943-23
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Cancer; Neoplasms; Bladder; Urothelial Tract
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms | interventions — larotaxel; Gemcitabine; Cisplatin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: larotaxel (XRP9881); Drug: cisplatin
- 2 (Active Comparator)
  Interventions: Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: larotaxel (XRP9881) — administered on day 1 as a 1-hour infusion
  Arms: 1
Drug: gemcitabine — administered on day 1, 8 and 15 as a 30-minute infusion
  Arms: 2
Drug: cisplatin — 1 hour infusion administered on day 1, 30 minutes after the other treatment

SUMMARY:
This is a randomized, open-label, multi-center study comparing the efficacy and safety of XRP9881 plus cisplatin to gemcitabine plus cisplatin in the first line treatment of locally advanced/metastatic urothelial tract or bladder cancer. The primary objective is to compare overall survival. Secondary objectives include comparisons of progression free survival, objective response rate, time to definitive deterioration of performance status, duration of response, time to definitive weight loss, and assessments of overall safety, and pharmacokinetics. Patients are treated until disease progression, death, or unacceptable toxicity and are followed-up until death or the end of the study whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histology/cytology confirmed Transitional Cell Carcinoma (TCC) with locally advanced (T4b) or metastatic urothelial tract or bladder cancer
* ECOG Performance Status 0 or 1
* No prior palliative chemotherapy

Exclusion Criteria:

* (Neo)Adjuvant chemotherapy if < 6 months between end of (neo)adjuvant chemotherapy and relapse
* Less than 6 weeks elapsed from prior radiotherapy and less than 3 weeks from surgery to time of randomization
* Prior cisplatin as (neo)adjuvant chemotherapy with cumulative dose > 300 mg/m²

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall survival defined as the time interval from the date of randomization to the date of death due to any cause | study period

SECONDARY OUTCOMES:
Radiological tumor assessments (CT/MRI) | at screening, every 8 weeks during treatment, at end of treatment, and in follow-up until documented disease progression
Adverse Events, laboratory assessments, vital signs, Physical Examinations, and ECOG Performance Status | at screening and every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (160):
- United States (52):
  - Sanofi-Aventis Investigational Site Number 840068, Anchorage, Alaska
  - Sanofi-Aventis Investigational Site Number 840035, Berkeley, California
  - Sanofi-Aventis Investigational Site Number 840012, Burbank, California
  - Sanofi-Aventis Investigational Site Number 840029, La Jolla, California
  - Sanofi-Aventis Investigational Site Number 840046, Los Angeles, California
  - Sanofi-Aventis Investigational Site Number 840003, Sacramento, California
  - Sanofi-Aventis Investigational Site Number 840005, San Bernardino, California
  - Sanofi-Aventis Investigational Site Number 840033, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840031, Denver, Colorado
  - Sanofi-Aventis Investigational Site Number 840032, Stamford, Connecticut
  - Sanofi-Aventis Investigational Site Number 840034, Washington D.C., District of Columbia
  - Sanofi-Aventis Investigational Site Number 840021, Washington D.C., District of Columbia
  - Sanofi-Aventis Investigational Site Number 840001, Boca Raton, Florida
  - Sanofi-Aventis Investigational Site Number 840048, Boynton Beach, Florida
  - Sanofi-Aventis Investigational Site Number 840049, Jacksonville, Florida
  - Sanofi-Aventis Investigational Site Number 840061, Lakeland, Florida
  - Sanofi-Aventis Investigational Site Number 840060, Athens, Georgia
  - Sanofi-Aventis Investigational Site Number 840030, Boise, Idaho
  - Sanofi-Aventis Investigational Site Number 840024, Maywood, Illinois
  - Sanofi-Aventis Investigational Site Number 840062, Peoria, Illinois
  - Sanofi-Aventis Investigational Site Number 840039, Goshen, Indiana
  - Sanofi-Aventis Investigational Site Number 840054, Kansas City, Kansas
  - Sanofi-Aventis Investigational Site Number 840057, Paducah, Kentucky
  - Sanofi-Aventis Investigational Site Number 840004, Metarie, Louisiana
  - Sanofi-Aventis Investigational Site Number 840045, Baltimore, Maryland
  - Sanofi-Aventis Investigational Site Number 840006, Detroit, Michigan
  - Sanofi-Aventis Investigational Site Number 840026, Lansing, Michigan
  - Sanofi-Aventis Investigational Site Number 840047, Saint Joseph, Michigan
  - Sanofi-Aventis Investigational Site Number 840009, Hackensack, New Jersey
  - Sanofi-Aventis Investigational Site Number 840044, Lake Success, New York
  - Sanofi-Aventis Investigational Site Number 840013, New York, New York
  - Sanofi-Aventis Investigational Site Number 840050, New York, New York
  - Sanofi-Aventis Investigational Site Number 840056, Rochester, New York
  - Sanofi-Aventis Investigational Site Number 840015, Syracuse, New York
  - Sanofi-Aventis Investigational Site Number 840041, Chapel Hill, North Carolina
  - Sanofi-Aventis Investigational Site Number 840007, Charlotte, North Carolina
  - Sanofi-Aventis Investigational Site Number 840019, Sylvania, Ohio
  - Sanofi-Aventis Investigational Site Number 840020, Bethlehem, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840065, Dunmore, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840058, Woonsocket, Rhode Island
  - Sanofi-Aventis Investigational Site Number 840052, Charleston, South Carolina
  - Sanofi-Aventis Investigational Site Number 840002, Knoxville, Tennessee
  - Sanofi-Aventis Investigational Site Number 840008, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840018, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840017, Lubbock, Texas
  - Sanofi-Aventis Investigational Site Number 840016, San Antonio, Texas
  - Sanofi-Aventis Investigational Site Number 840064, Temple, Texas
  - Sanofi-Aventis Investigational Site Number 840010, The Woodlands, Texas
  - Sanofi-Aventis Investigational Site Number 840036, Seattle, Washington
  - Sanofi-Aventis Investigational Site Number 840011, Madison, Wisconsin
  - Sanofi-Aventis Investigational Site Number 840025, Marshfield, Wisconsin
  - Sanofi-Aventis Investigational Site Number 840038, Milwaukee, Wisconsin
- Argentina (5):
  - Sanofi-Aventis Investigational Site Number 032002, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032003, Ciudad de Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032004, Mendoza
  - Sanofi-Aventis Investigational Site Number 032005, Rosario
  - Sanofi-Aventis Investigational Site Number 032001, Santa Fe
- Australia (3):
  - Sanofi-Aventis Investigational Site Number 036002, Adelaide
  - Sanofi-Aventis Investigational Site Number 036003, Bedford Park
  - Sanofi-Aventis Investigational Site Number 036004, St Leonards
- Belgium (6):
  - Sanofi-Aventis Investigational Site Number 056005, Aalst
  - Sanofi-Aventis Investigational Site Number 056001, Brussels
  - Sanofi-Aventis Investigational Site Number 056002, Brussels
  - Sanofi-Aventis Investigational Site Number 056004, Ottignies
  - Sanofi-Aventis Investigational Site Number 056003, Wilrijk
  - Sanofi-Aventis Investigational Site Number 056006, Yvoir
- Brazil (7):
  - Sanofi-Aventis Investigational Site Number 076006, Barretos
  - Sanofi-Aventis Investigational Site Number 076004, Florianópolis
  - Sanofi-Aventis Investigational Site Number 076001, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076003, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076002, Rio de Janeiro
  - Sanofi-Aventis Investigational Site Number 076007, São Paulo
  - Sanofi-Aventis Investigational Site Number 076005, São Paulo
- Canada (5):
  - Sanofi-Aventis Investigational Site Number 124007, Edmonton
  - Sanofi-Aventis Investigational Site Number 124001, London
  - Sanofi-Aventis Investigational Site Number 124006, Montreal
  - Sanofi-Aventis Investigational Site Number 124003, Québec
  - Sanofi-Aventis Investigational Site Number 124002, Weston
- Sanofi-Aventis Investigational Site Number 152001, Santiago, Chile
- France (10):
  - Sanofi-Aventis Investigational Site Number 250006, Avignon
  - Sanofi-Aventis Investigational Site Number 250003, Bordeaux
  - Sanofi-Aventis Investigational Site Number 250005, Hyères
  - Sanofi-Aventis Investigational Site Number 250011, Le Mans
  - Sanofi-Aventis Investigational Site Number 250004, Lyon
  - Sanofi-Aventis Investigational Site Number 250012, Perpignan
  - Sanofi-Aventis Investigational Site Number 250007, Poitiers
  - Sanofi-Aventis Investigational Site Number 250008, Saint-Herblain
  - Sanofi-Aventis Investigational Site Number 250009, Strasbourg
  - Sanofi-Aventis Investigational Site Number 250001, Suresnes
- India (6):
  - Sanofi-Aventis Investigational Site Number 356003, Bangalore
  - Sanofi-Aventis Investigational Site Number 356007, Kolkata
  - Sanofi-Aventis Investigational Site Number 356004, New Delhi
  - Sanofi-Aventis Investigational Site Number 356001, New Delhi
  - Sanofi-Aventis Investigational Site Number 356002, Vellore
  - Sanofi-Aventis Investigational Site Number 356005, Visakhapatnam
- Israel (6):
  - Sanofi-Aventis Investigational Site Number 376005, Haifa
  - Sanofi-Aventis Investigational Site Number 376004, Kfar Saba
  - Sanofi-Aventis Investigational Site Number 376003, Petah Tikva
  - Sanofi-Aventis Investigational Site Number 376002, Tel Aviv
  - Sanofi-Aventis Investigational Site Number 376007, Tel Litwinsky
  - Sanofi-Aventis Investigational Site Number 376001, Tzrifin
- Italy (7):
  - Sanofi-Aventis Investigational Site Number 380004, Bari
  - Sanofi-Aventis Investigational Site Number 380003, Lecce
  - Sanofi-Aventis Investigational Site Number 380005, Meldola
  - Sanofi-Aventis Investigational Site Number 380006, Pavia
  - Sanofi-Aventis Investigational Site Number 380002, Perugia
  - Sanofi-Aventis Investigational Site Number 380001, Roma
  - Sanofi-Aventis Investigational Site Number 380008, Viterbo
- Mexico (4):
  - Sanofi-Aventis Investigational Site Number 484003, Aguascalientes
  - Sanofi-Aventis Investigational Site Number 484007, Chihuahua City
  - Sanofi-Aventis Investigational Site Number 484005, Chihuahua City
  - Sanofi-Aventis Investigational Site Number 484004, Monterrey
- Netherlands (7):
  - Sanofi-Aventis Investigational Site Number 528005, Amsterdam
  - Sanofi-Aventis Investigational Site Number 528002, Arnhem
  - Sanofi-Aventis Investigational Site Number 528006, Hoofddorp
  - Sanofi-Aventis Investigational Site Number 528003, Maastricht
  - Sanofi-Aventis Investigational Site Number 528004, Nijmegen
  - Sanofi-Aventis Investigational Site Number 528001, Sittard-Geleen
  - Sanofi-Aventis Investigational Site Number 528007, Zwolle
- Poland (4):
  - Sanofi-Aventis Investigational Site Number 616002, Poznan
  - Sanofi-Aventis Investigational Site Number 616004, Rybnik
  - Sanofi-Aventis Investigational Site Number 616001, Warsaw
  - Sanofi-Aventis Investigational Site Number 616005, Wroclaw
- Russia (11):
  - Sanofi-Aventis Investigational Site Number 643009, Chelyabinsk
  - Sanofi-Aventis Investigational Site Number 643010, Kursk
  - Sanofi-Aventis Investigational Site Number 643006, Moscow
  - Sanofi-Aventis Investigational Site Number 643008, Moscow
  - Sanofi-Aventis Investigational Site Number 643004, Moscow
  - Sanofi-Aventis Investigational Site Number 643005, Moscow
  - Sanofi-Aventis Investigational Site Number 643001, Obninsk
  - Sanofi-Aventis Investigational Site Number 643002, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643003, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643007, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643011, Saint Petersburg
- South Africa (7):
  - Sanofi-Aventis Investigational Site Number 710008, Bloemfontein
  - Sanofi-Aventis Investigational Site Number 710003, Cape Town
  - Sanofi-Aventis Investigational Site Number 710001, Cape Town
  - Sanofi-Aventis Investigational Site Number 710007, Durban
  - Sanofi-Aventis Investigational Site Number 710009, Durban
  - Sanofi-Aventis Investigational Site Number 710006, Port Elizabeth
  - Sanofi-Aventis Investigational Site Number 710005, Pretoria
- Spain (12):
  - Sanofi-Aventis Investigational Site Number 724006, Badalona
  - Sanofi-Aventis Investigational Site Number 724001, Barcelona
  - Sanofi-Aventis Investigational Site Number 724004, Barcelona
  - Sanofi-Aventis Investigational Site Number 724008, Barcelona
  - Sanofi-Aventis Investigational Site Number 724002, Barcelona
  - Sanofi-Aventis Investigational Site Number 724003, Madrid
  - Sanofi-Aventis Investigational Site Number 724010, Oviedo
  - Sanofi-Aventis Investigational Site Number 724013, Palma de Mallorca
  - Sanofi-Aventis Investigational Site Number 724007, Palma de Mallorca
  - Sanofi-Aventis Investigational Site Number 724009, Pamplona
  - Sanofi-Aventis Investigational Site Number 724011, Santiago de Compostela
  - Sanofi-Aventis Investigational Site Number 724012, Zaragoza
- Sweden (2):
  - Sanofi-Aventis Investigational Site Number 752001, Umeå
  - Sanofi-Aventis Investigational Site Number 752002, Uppsala
- Turkey (Türkiye) (5):
  - Sanofi-Aventis Investigational Site Number 792002, Ankara
  - Sanofi-Aventis Investigational Site Number 792003, Ankara
  - Sanofi-Aventis Investigational Site Number 792004, Ankara
  - Sanofi-Aventis Investigational Site Number 792006, Istanbul
  - Sanofi-Aventis Investigational Site Number 792001, Istanbul